CLINICAL TRIAL: NCT00831493
Title: Phase I/II Trial of Vorinostat and Radiation Therapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Vorinostat Plus Radiation Therapy in Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0780
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Pancreatic Cancer; Locally Advanced Pancreatic Cancer; LAPC; Non-Metastatic; Unresectable; Vorinostat; XRT; RT; Radiation Therapy; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Chemoradiotherapy; Radiotherapy; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat + Radiation Therapy (Experimental): Vorinostat starting dose 200 mg orally once daily, Monday to Friday, Weeks 1 to 6; Radiation Therapy Dose of 50.4 Gray (Gy) in 1.8 Gy fractions in 28 fractions, Monday to Friday, Weeks 1 to 6.
  Interventions: Radiation: Chemoradiation (Radiation Therapy); Drug: Vorinostat

INTERVENTIONS:
Radiation: Chemoradiation (Radiation Therapy) — Dose of 50.4 Gy in 1.8 Gy fractions in 28 fractions, Monday to Friday, Weeks 1 to 6.
  Other Names: XRT; RT
Drug: Vorinostat — Starting Dose of 200 mg orally once daily, Monday to Friday, Weeks 1 to 6.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390

SUMMARY:
Primary Endpoint:

To determine the maximum tolerated dose (MTD) of vorinostat + radiation therapy (RT) in patients with locally advanced pancreatic cancer (LAPC).

Secondary Endpoints:

1. To assess the efficacy of vorinostat + RT in patients with LAPC as estimated by median overall survival.
2. To determine the radiological response as assessed by regular computer tomography (CT) and/or dynamic contrast enhanced computer tomography (DCE-CT) among patients treated with vorinostat and RT.
3. To evaluate the occurrence of symptoms and correlate to disease progression and tolerance to treatment using the MD Anderson Symptom Inventory-Gastrointestinal Module (MDASI-GI) self-reporting tool.
4. To correlate serum cytokine levels with symptoms and treatment outcomes.

DETAILED DESCRIPTION:
The Study Drugs:

Vorinostat is designed to interfere with the growth of cancer cells.

Study Drug Dose Level:

If you are found to be eligible to take part in the study, you will begin receiving vorinostat. The dose you receive will be based on how many participants have been enrolled before you, and on the safety data available. The first group of 3 enrolled participants will be given low doses of vorinostat. If no intolerable side effects occur, the next group of 3 will be enrolled at a higher dose level. The study doctor will tell you what dose you will be receiving and how it compares to the doses other participants have received. Up to 3 dose levels will be tested.

Study Drug Administration:

On each day that you receive radiation, you will take vorinostat (as a capsule taken by mouth) in the morning with food.

Radiation:

You will receive radiation once a day on Monday through Friday, except for holidays. This schedule will be continued for 5 1/2 weeks or 28 doses total. Each radiation treatment will usually last about 10-15 minutes.

Surgical Evaluation:

After completing radiation therapy, you will come back for a follow-up visit about 6-12 weeks later.

Length of Study:

You will remain on study for up to 5 1/2 weeks. You will be taken off-study early if the disease gets worse or intolerable side effects occur.

This is an investigational study. Vorinostat is FDA approved and commercially available. The use of vorinostat for pancreatic cancer and in combination with radiation is investigational. At this time, this combination is being used in research only.

Up to 37 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
2. Patients must be >/= 18 years of age. There will be no upper age restriction.
3. Cytologic or histologic proof of adenocarcinoma of the pancreas. Patients can have tumor originating in any part of the pancreas. Islet cell tumors are not eligible. Only patients with non- metastatic, unresectable disease (American Joint Committee on Cancer (AJCC) 2002 stage T4 NX M0) are eligible. Patients who cannot undergo resection because of underlying medical problems are also eligible. Patients with regional nodal disease are eligible.
4. All patients must be staged with a physical exam, chest x-ray/CXR, and contrast-enhanced helical thin-cut abdominal CT. Unresectability is defined by CT criteria: a) evidence of tumor extension to the celiac axis or superior mesenteric (SM) artery, or b) evidence on either CT or angiogram of occlusion of the SM vein or SM/ portal vein confluence. If a tumor does not meet this definition and is found to be unresectable at surgical exploration, then that tumor is considered unresectable.
5. Patients may have received prior chemotherapy but not prior radiation therapy to the upper abdomen.
6. Bone marrow function: absolute neutrophil count (ANC) >1,500/ul. Platelets >100,000/ul.
7. Hepatic function: Total bilirubin less than 1.5mg/dL. If the patient required an endobiliary stent and/or external biliary drain, the bilirubin level must have declined on consecutive measurements indicating adequate biliary decompression; alanine aminotransferase (ALT) </= 5 times the upper limit of normal.
8. Renal function: Blood urea nitrogen (BUN) </= 30 mg% and creatinine </= 1.5 mg%
9. Patients must be willing to sign informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary.

Exclusion Criteria:

1. Prior abdominal radiotherapy.
2. Participation in any other experimental drug study in the 30 days preceding initiation of treatment on the current study.
3. Prior treatment with HDAC inhibitors (except valproic acid with a 30-day washout period)
4. Prior history of cancer within the last five years except for basal cell carcinoma of the skin or carcinoma in situ of the cervix. Patients with previous malignancies but without evidence of disease for 5 years will be allowed to enter the trial.
5. Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Women / men of childbearing potential not using a reliable contraceptive method (oral contraceptive, other hormonal contraceptive, intrauterine device, diaphragm or condom). (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential). Patients must agree to continue contraception for 30 days from the date of the last study drug administration.
6. Serious, uncontrolled, concurrent infection(s) requiring intravenous (IV) antibiotics or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
7. Current treatment of active hepatitis virus or HIV infection with interferon, ribavirin, telbivudine, entecavir, lamivudine, adefovir, efavirenz, zidovudine, tenofovir, emtricitabine, or ritonavir.
8. Psychiatric disorders rendering patients incapable of complying with the requirements of the protocol.
9. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Krishnan, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period is May 8, 2009 to October 5, 2010. All participants were recruited at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Vorinostat + Radiation Therapy
Started | 3
Completed | 2
Not Completed | 1
Not completed — Intractable nausea and vomiting | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat + Radiation Therapy
Number analyzed (Participants) | 3
Age Continuous [Median (Full Range); unit: years] | 55 [40 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vorinostat + Chemoradiation
Description: MTD is maximum dose at which 6 patients are treated and there is at most 1 patient with dose limiting toxicities (DLT). Toxicities graded according to the Common Terminology Criteria for Adverse events (CTCAE).
Time Frame: Toxicity assessment at 6 weeks following chemoradiation (6 weeks)
Population: Analysis per protocol; Of the three participants enrolled only two were eligible for MTD calculation.
Measure: Number; unit: mg
Arm/Group | Vorinostat + Radiation Therapy
Number analyzed (Participants) | 2
mg | 200

ADVERSE EVENTS:
Time Frame: 2.5 months
Arm/Group | Vorinostat + Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat + Radiation Therapy (N=3)
vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No